CLINICAL TRIAL: NCT05310877
Title: Feasibility and Acceptability of a Values-Affirmation Intervention Targeting Medication Adherence in Older Adults With Heart Failure
Brief Title: Values-Affirmation Intervention Targeting Medication Adherence in Older Adults With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5K23AG061214 (NIH); 5K23AG061214 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-04-05 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Values-affirmation (Experimental)
  Interventions: Behavioral: Values-Affirmation

INTERVENTIONS:
Behavioral: Values-Affirmation — Participants will engage in a brief values-affirmation exercise to target personal motivation and openness to medication adherence. The interventionist will then review tailored medication education and individual skills training recommendations. Following the intervention session, participants will receive electronic pill box(es) that are labeled with the participants' most important core value(s) and will be asked to use these pill box(es) to take their HF medications for 4 weeks.

SUMMARY:
Heart failure (HF) represents a significant public health concern. Medication non-adherence represents a modifiable contributor to costly hospital readmissions in older adults with HF. Educational interventions improve, but do not eliminate, non-adherence. Values affirmation interventions which invite individuals to reflect on core values may encourage better engagement in health behaviors by increasing the personal relevance of targeted behaviors. Similar interventions have promoted weight loss, increased adherence and physical activity, and more frequent fruit and vegetable consumption in a variety of contexts and populations. This study seeks to test a recently developed values-affirmation intervention targeting medication adherence in older adults with HF enrolled in cardiac rehabilitation (CR). The purpose of this feasibility study is to test methodology to aid development of a subsequent randomized controlled pilot trial to examine preliminary efficacy.

DETAILED DESCRIPTION:
The objective of this study is to examine the preliminary feasibility and acceptability of study procedures and the values-affirmation intervention in a single-arm trial. Participants will be asked to complete a brief intervention with tailored education relevant to medication information, motivation, and behavioral skills. Participants will complete a baseline assessment and a follow-up assessment at one month post-intervention. The investigators hypothesize that the developed study and intervention procedures will be feasible and acceptable to participants. The investigators will also examine changes in self-reported and electronically monitored medication adherence from the baseline assessment to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure
* Enrolled in cardiac rehabilitation
* Read and understand English
* At risk for medication non-adherence based on self-report screening or number of prescribed medications

Exclusion Criteria:

* Current participation in another medication-monitoring clinical or research protocol
* New York Heart Association class IV heart failure
* Diagnosis of Alzheimer's, dementia, or severe cognitive impairment indicated on screening
* Current suicidality or psychosis
* Terminal illness with an expected lifespan of less than 6 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Values-affirmation
Started | 7
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Values-affirmation
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data for 1 participant on age
  years
    number analyzed (Participants) | 6
    (all) | 75.5 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment Procedures
Description: Proportion of eligible participants who enroll in the study
Time Frame: Baseline
Population: Number of participants who completed eligibility screening and met all study criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Values-affirmation
Number analyzed (Participants) | 10
Participants | 7

2. Primary Outcome: Feasibility of Intervention Procedures
Description: Proportion of enrolled participants who complete the study
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Values-affirmation
Number analyzed (Participants) | 7
Participants | 6

3. Primary Outcome: Acceptability Assessed Via Qualitative Exit Interview- Number of Participants Who Completed Interview
Description: Qualitative exit interview to assess patient reported satisfaction with intervention content, intervention delivery, and study procedures
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Values-affirmation
Number analyzed (Participants) | 7
Participants | 7

4. Secondary Outcome: Self-reported Medication Adherence
Description: Timeline follow-back interview
Time Frame: Baseline, 4 weeks
Population: At 4 weeks, 2 participants refused to complete EOT survey
Measure: Mean (Standard Deviation); unit: percent adherence
Arm/Group | Values-affirmation
Number analyzed (Participants) | 7
percent adherence
  Baseline | 96.69 (3.82)
  4 weeks: number analyzed (Participants) | 5
  4 weeks | 99.05 (2.13)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Values-affirmation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Values-affirmation (N=7)
Chest pain- cardiac (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Values-affirmation (N=7)
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/77/NCT05310877/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/77/NCT05310877/SAP_001.pdf